CLINICAL TRIAL: NCT02391896
Title: Design and Evaluation of Innovative Mobile X-Ray Technology for Rapid and Accurate Diagnosis of Thoracic Disease in Critically Ill Patients
Brief Title: Design and Evaluation of Mobile X-ray for Rapid and Accurate Diagnosis of Thoracic Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has left UHN. This study is no longer running at UHN.
Sponsor: University Health Network, Toronto (Other)
Collaborators: Carestream Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 14-7549-CE
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Thoracic Diseases
MeSH Terms: conditions — Thoracic Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Digital Tomosynthesis (Other): Patient will get tomosynthesis scan
  Interventions: Device: Dual energy and tomosynthesis xray
- Dual energy (Other): Patient will get dual energy scan
  Interventions: Device: Dual energy and tomosynthesis xray

INTERVENTIONS:
Device: Dual energy and tomosynthesis xray

SUMMARY:
Computed tomography (CT) is the most accurate test for evaluating patients with thoracic disease. However, access to CT is limited due to long wait times and for the sickest patients in Hospital who cannot be transported from the ward to the CT scanner. The investigators propose to modify a standard X-ray unit to provide more detailed information of the chest such that a CT scan is not required for all patients.

DETAILED DESCRIPTION:
Dual-energy (DE) imaging consists of acquiring paired "low" and "high"-energy x-ray images. The use of DE to improve radiological contrast was first described by Jacobson et al in 1958; followed by Mistretta et al and Alvarez and Macovski in the mid-1970s. With the advent of new digital X-ray detectors that provide high dose efficiency and rapid readout of digital X-ray projections, there has been renewed interest in using DE x-ray imaging for lung nodule detection. More recently, portable x-ray detectors have made bedside DE imaging possible. Jabri et. al. presented a portable DE system with novel respiratory and cardiac gating, and Hoggarth et. al. investigated the potential for DE subtraction in improving the visualization of lung tumors while performing image-guided radiotherapy.

The investigators group is experienced in investigating DE for lung nodule detection, this theoretical framework was instrumental in optimizing a clinical prototype for high-performance DE chest X-ray. It identified optimal DE image acquisition and decomposition techniques, and validated the approach in comparison to human observer performance. The analysis further demonstrated that - given a high-performance flat plate detector, optimal acquisition and decomposition - DE chest X-ray is possible at the same dose as conventional computer radiography (CR) and digital radiography (DR) chest X-ray, while significantly improving conspicuity of subtle lung nodules by the reduction of overlying background noise. The DE work undertaken by our group is unique in terms of providing a clear theoretical framework for optimizing a clinical prototype for best performance in terms of image quality and patient exposure to ionizing radiation.

ELIGIBILITY:
Inclusion Criteria:

* the presence of lung disease (nodules, masses, consolidation and collapse), pleural disease (effusion, thickening), mediastinal and hilar lymph node enlargement, on thoracic CT

Exclusion Criteria:

* unable to consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Improved detection of maliganancy with modified x-ray | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Narinder Paul, MD, Principal Investigator — UHN
Locations (1):
- Toronto General Hospital, Department of Medical Imaging, Toronto, Ontario, Canada